CLINICAL TRIAL: NCT00329641
Title: Phase II Trial of BAY 43-9006 (Sorafenib; NSC-724772) in Combination With Carboplatin and Paclitaxel in Patients With Metastatic Uveal Melanoma
Brief Title: Sorafenib, Carboplatin, and Paclitaxel in Treating Patients With Stage IV Melanoma of the Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00777; NCI-2009-00777 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000467188; S0512; S0512 (Other: Southwest Oncology Group); S0512 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Results first posted 2012-07-11 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2013-10

CONDITIONS: Ciliary Body and Choroid Melanoma, Medium/Large Size; Extraocular Extension Melanoma; Iris Melanoma; Metastatic Intraocular Melanoma; Recurrent Intraocular Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Carboplatin; Paclitaxel; Sorafenib

ARMS (1):
- Treatment (carboplatin, paclitaxel, sorafenib) (Experimental): Patients receive carboplatin IV and paclitaxel IV once on day 1 and oral sorafenib twice daily on days 2-19. Treatment repeats every 21 days for up to 6 courses.* After 6 courses, patients continue to receive oral sorafenib alone twice daily in the absence of disease progression or unacceptable toxicity.
  [Note: *If sorafenib is discontinued prior to course 6, patients may continue to receive carboplatin and paclitaxel for up to 6 courses; if carboplatin and paclitaxel are discontinued prior to course 6, patients may continue to receive sorafenib alone twice daily on days 1-21 of each course in the absence of disease progression or unacceptable toxicity. ]
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: paclitaxel — Given IV
Drug: sorafenib tosylate — Given orally

SUMMARY:
This phase II trial is studying how well sorafenib works when given together with carboplatin and paclitaxel in treating patients with stage IV melanoma of the eye. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib may help carboplatin and paclitaxel work better by making tumor cells more sensitive to the drugs. Sorafenib may also stop the growth of melanoma by blocking some of the enzymes needed for tumor cell growth and by blocking blood flow to the tumor. Giving sorafenib together with carboplatin and paclitaxel may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate (confirmed and unconfirmed, complete and partial response) of patients with stage IV uveal melanoma treated with sorafenib, carboplatin, and paclitaxel.

SECONDARY OBJECTIVES:

I. Determine the overall and progression-free survival of patients treated with this regimen.

II. Determine the toxic effects of this regimen in these patients. III. Determine, preliminarily, the relationship between clinical outcomes and baseline microvessel density (MVD) in tumor specimens, changes in vascular endothelial growth factor (VEGF) levels in plasma and urine, changes in MVD, changes in VEGF receptor-2 phosphorylation in tumor, and/or changes in ERK 1/2 phosphorylation in stimulated lymphocytes and tumor.

OUTLINE: This is a non-randomized, open-label, multicenter study.

Patients receive carboplatin IV and paclitaxel IV once on day 1 and oral sorafenib twice daily on days 2-19. Treatment repeats every 21 days for up to 6 courses.* After 6 courses, patients continue to receive oral sorafenib alone twice daily in the absence of disease progression or unacceptable toxicity.

[Note: *If sorafenib is discontinued prior to course 6, patients may continue to receive carboplatin and paclitaxel for up to 6 courses; if carboplatin and paclitaxel are discontinued prior to course 6, patients may continue to receive sorafenib alone twice daily on days 1-21 of each course in the absence of disease progression or unacceptable toxicity. ]

After completion of study treatment, patients are followed periodically for up to 3 years.

ELIGIBILITY:
Criteria:

* Histologically proven uveal melanoma
* Must have documented disease progression during or after =< 1 prior systemic treatment
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan
* No tumor involving major vessels
* Zubrod performance status 0-1
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine =< 2 times upper limit of normal (ULN)
* Bilirubin =< 2 times ULN
* SGOT or SGPT =< 2 times ULN (5 times ULN if hepatic metastasis present)
* INR in range (usually between 2 and 3)
* No active bleeding
* No bleeding diathesis, active coagulopathy, or pathological condition that carries a high risk of bleeding
* No condition (e.g., gastrointestinal tract disease) affecting ability to take oral medication or requiring IV alimentation
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer for which the patient is currently in complete remission, or any other cancer for which the patient has been disease-free for 5 years
* At least 28 days since prior systemic treatment for this disease comprising 1 of the following: single chemotherapy agent/regimen; single immunotherapy agent/regimen; single investigational treatment agent/regimen
* At least 21 days since prior major surgery
* No prior sorafenib or any other agents targeting raf kinase or vascular endothelial growth factor (VEGF) or VEGF receptor
* No prior surgical procedures affecting absorption
* No concurrent systemic corticosteroid therapy
* Topical and/or inhaled steroids are allowed
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, and phenobarbital), rifampin, or Hypericum perforatum (St. John's wort)
* No prophylactic granulocyte/platelet colony-stimulating factors during the first course of treatment
* Concurrent full-dose oral anticoagulants (e.g., warfarin) are allowed provided all of the following criteria are met: in-range INR ; stable dose of oral anticoagulant; no active bleeding or high risk of bleeding
* Stage IV disease
* No known varices
* No uncontrolled hypertension with systolic blood pressure (BP) > 140 mm Hg or diastolic BP > 90 mm Hg
* No significant traumatic injury within the past 21 days
* No active, uncontrolled peptic ulcer disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Aparicio, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States

REFERENCES:
- [Derived] Bhatia S, Moon J, Margolin KA, Weber JS, Lao CD, Othus M, Aparicio AM, Ribas A, Sondak VK. Phase II trial of sorafenib in combination with carboplatin and paclitaxel in patients with metastatic uveal melanoma: SWOG S0512. PLoS One. 2012;7(11):e48787. doi: 10.1371/journal.pone.0048787. Epub 2012 Nov 30. PMID 23226204

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib, Carboplatin, Paclitaxel: Standard carboplatin and paclitaxel doses with the addition of sorafenib (800 mg daily)
Period: Overall Study
Arm/Group | Sorafenib, Carboplatin, Paclitaxel
Started | 25
Eligible | 25
Eligible and Received Treatment | 24
Completed | 19
Not Completed | 6
Not completed — Did not start treatment | 1
Not completed — Not eligible | 1
Not completed — Adverse Event | 3
Not completed — Other reason, not protocol specified | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib, Carboplatin, Paclitaxel
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: Years] | 61 [48 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial Response)
Description: Complete response corresponds to complete disappearance of all measurable and non-measurable lesions with no new lesions. Partial response corresponds to greater than or equal to 30ﬁ decrease of sum of longest diameter of all target measurable lesions with no new lesion and non unequivocal progression of non-measurable disease.
Time Frame: Every 6 weeks for the first 8 cycles of therapy, then every three cycles (9 weeks) until progression
Population: Eligible patients who received some treatment
Measure: Number; unit: participants
Arm/Group | Sorafenib, Carboplatin, Paclitaxel
Number analyzed (Participants) | 24
participants | 0

2. Secondary Outcome: One-year Overall Survival
Description: Measured from date of registration to study until death due to any caused with observations last known to be alive censored at the date of last contact
Time Frame: Every 6-9 weeks until progression, after progression every six months for first two years and annually thereafter up to 3 for up to 3 years after registration or until death
Population: Eligible patients who received some treatment
Measure: Number (95% Confidence Interval); unit: Percentage of population
Arm/Group | Sorafenib, Carboplatin, Paclitaxel
Number analyzed (Participants) | 24
Percentage of population | 42 [22 to 60]

3. Secondary Outcome: 6-month Progression-free Survival
Description: Measured from the date of registration to the first of progression or death due to any cause with patients last known to be alive and progression-free censored at the date of last contact
Time Frame: Every 6 weeks for the first 8 cycles of therapy, and then every 9 weeks until disease progression for up to 3 years after registration or until death
Measure: Number (95% Confidence Interval); unit: Percent of population
Arm/Group | Sorafenib, Carboplatin, Paclitaxel
Number analyzed (Participants) | 24
Percent of population | 29 [13 to 48]

4. Secondary Outcome: Toxicity
Description: Number of patients with Grade 3-5 adverse events that are related to study drug by given type of adverse event
Time Frame: Weekly during the first cycle of therapy, then prior to each cycle (one cycle = 3 weeks)
Population: Eligible patients who started therapy
Measure: Number; unit: Participants with a given type of AE
Groups:
- Intervention: Sorafenib, Carboplatin, Paclitaxel
Arm/Group | Intervention
Number analyzed (Participants) | 24
Participants with a given type of AE
  Calcium, serum-low (hypocalcemia) | 1
  Cataract | 1
  Diarrhea | 2
  Fatigue (asthenia, lethargy, malaise) | 1
  Febrile neutropenia | 1
  Hemoglobin | 2
  Infec w/ Gr 3/4 neut-Urinary tract | 1
  Leukocytes (total WBC) | 4
  Lymphopenia | 2
  Mucositis/stomatitis (func/symp) - Pharynx | 1
  Neuropathy: sensory | 2
  Neutrophils/granulocytes (ANC/AGC) | 10
  Platelets | 4
  Pruritus/itching | 1
  Rash/desquamation | 5
  Vision-blurred vision | 1

ADVERSE EVENTS:
Time Frame: While the patient is on treatment until resolution of acute toxicities with maximum grade reported
Description: Regular investigator assessments are reported after each cycle of protocol treatment
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 2/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=24)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=24)
Hemoglobin (Blood and lymphatic system disorders) | 5
Vision-blurred vision (Eye disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 11
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 2
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Edema: limb (General disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2
Leukocytes (total WBC) (Investigations) | 7
Lymphopenia (Investigations) | 4
Metabolic/Laboratory-Other (Specify) (Investigations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 10
Platelets (Investigations) | 7
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 7
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3
Pain - Joint (Musculoskeletal and connective tissue disorders) | 4
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 6
Neuropathy: motor (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 19
Taste alteration (dysgeusia) (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 2
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 3
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 10
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less